CLINICAL TRIAL: NCT01186458
Title: A Phase II Study of Fludarabine, Velcade and Rituximab for Relapsed or Refractory Follicular Non-Hodgkin Lymphoma: Hoosier Oncology Group LYM08-134
Brief Title: Fludarabine, Velcade and Rituximab for Relapsed or Refractory Follicular Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: Genentech, Inc. (Industry); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOG LYM08-134
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-08

CONDITIONS: Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — fludarabine; Bortezomib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fludarabine, Velcade and Rituximab (Experimental): Fludarabine, Velcade and Rituximab
  Interventions: Drug: Fludarabine; Drug: Velcade; Drug: Rituximab

INTERVENTIONS:
Drug: Fludarabine — Fludarabine 25 mg/m2 IV over 30 minutes on days 1, 2, 4. Cycle = 28 days; maximum of 6 cycles of therapy.
Drug: Velcade — Velcade (given after fludarabine)1.3 mg/m2 IV push over 3 to 5 seconds on days 1, 4, 8, 11. Cycle = 28 days; maximum of 6 cycles of therapy.
Drug: Rituximab — Rituximab given after Velcade) 375 mg/m2 IV piggyback on day 1. Cycle = 28 days; maximum of 6 cycles of therapy.

SUMMARY:
The purpose of this study is to determine the effectiveness of fludarabine, Velcade, and rituximab treatment regimen in patients with relapsed or refractory follicular non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

* Fludarabine 25 mg/m2 IV over 30 minutes , Days 1, 2, 4
* Velcade(given after fludarabine) 1.3 mg/m2 IV push over 3 to 5 seconds, Days 1, 4, 8, 11
* Rituximab (given after Velcade) 375 mg/m2 IV piggyback, Day 1
* Cycle = 28 days; max 6 cycles

ECOG Performance Status: 0-2

Life Expectancy: Not specified

Hematopoietic:

* Absolute neutrophil count (ANC) ≥ 1.5 K/mm3 (ANC > 0.5 K/mm3 if known lymphomatous involvement of the bone marrow).
* Platelets ≥ 100 K/mm3 (Platelets >50 K/mm3 if known lymphomatous involvement of the bone marrow).

Hepatic:

* Total bilirubin ≤1.5 ULN
* Aspartate aminotransferase (AST, SGOT) ≤ 2.5 x ULN
* Alanine aminotransferase (ALT, SGPT) ≤ 2.5 x ULN

Renal:

* Creatinine < 1.5 x institutional upper limit (ULN) or creatinine clearance ≥ 50 cc/min

Cardiovascular:

* No myocardial infarction within 6 months prior to enrollment
* No heart failure per New York Heart Association Classification III or IV
* No severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically confirmed Follicular Non-Hodgkin Lymphoma (Grade I, II, or IIIa)
* Must have measurable disease defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded as ≥2 cm with conventional techniques or as >1 cm with spiral CT scan) and obtained by imaging within 30 days prior to registration for protocol therapy.
* Must have received at least one prior therapeutic regimen, but no more than three prior regimens of conventional cytotoxic therapy. NOTE: Prior recipients of stem cell transplantation will be included, with the preparative cytoreductive and high-dose therapies counted collectively as one prior therapy.
* Must be off all cytotoxic chemotherapy for at least four weeks prior to registration for protocol therapy (6 weeks for BCNU or mitomycin C).
* Patients are allowed to have received one course of prior radioimmunotherapy (RIT: either tositumomab or ibritumomab). NOTE: Radioimmunotherapy must be completed at least 12 weeks prior to registration for protocol therapy with recovery to baseline of ANC and platelets.
* Prior fludarabine, Velcade or rituximab is allowed as long as therapy is completed at least 30 days prior to registration for protocol therapy. Patients may be refractory (defined as not responding or demonstrating progressive disease in <6 months) to prior rituximab. Patients may not be refractory to prior fludarabine or Velcade.
* Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed and for 30 days following protocol therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to prior to registration for protocol therapy. NOTE: Patients are considered of child bearing potential unless they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal (no menses for at least 12 months).
* Females must not be breastfeeding.
* Males must agree to use an acceptable method of contraception for the duration of the study.

Exclusion Criteria:

* No current active CNS metastases. Patients with neurological symptoms must undergo a head CT scan or brain MRI to exclude brain metastasis within 7 days prior to registration for protocol therapy. NOTE: Patients with treated brain metastasis must be off steroids or on tapering or stable doses of steroids and have completed radiation at least 30 days prior to registration for protocol therapy.
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, Gleason ≤ grade 6 prostate cancers, or other cancer for which the subject has been disease-free for at least 3 years.
* No treatment with any investigational agent within 30 days prior to registration for protocol therapy.
* Prior radiation therapy is allowed to < 25% of the bone marrow. NOTE: No radiation therapy within 30 days prior to registration for protocol therapy.
* No clinically significant infections as judged by the treating investigator.
* No active HIV, hepatitis B or hepatitic C infection.
* No cerebrovascular accident (CVA) within 6 months of study enrollment.
* No psychiatric illness/social situations that would limit compliance with study requirements.
* No history of hypersensitivity to Velcade, boron or mannitol.
* No peripheral neuropathy grade > 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shivani Srivastava, M.D., Study Chair — Hoosier Cancer Research Network
Locations (11):
- United States (11):
  - Cancer Care Center of Southern Indiana, Bloomington, Indiana
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Community Regional Cancer Center, Indianapolis, Indiana
  - Arnett Cancer Care, Lafayette, Indiana
  - Virtua Health Cancer Program, Mount Holly, New Jersey
  - South Jersey Health Care, Vineland, New Jersey
  - University of Rochester Medical Center, Rochester, New York
  - Case Comprehensive Cancer Center - University Hospitals Case Medical Center, Cleveland, Ohio
  - Seidman Cancer Center, Cleveland, Ohio
  - Reading Hospital Regional Cancer Center, West Reading, Pennsylvania

REFERENCES:
- See also: Hoosier Oncology Group Homepage — http://www.hoosieroncologygroup.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fludarabine, Velcade and Rituximab
Started | 4
Completed | 3
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Fludarabine, Velcade and Rituximab
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.50 (14.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: To determine the overall response rate and frequency of complete and partial responses in patients with relapsed or refractory follicular non-Hodgkin lymphoma (NHL) who receive therapy with fludarabine, Velcade, and rituximab administered every 28 days.
Time Frame: 6 months
Population: Data for this primary objective was not collected or analyzed due to the termination of the study.
Arm/Group | Fludarabine, Velcade and Rituximab
Number analyzed (Participants) | 0

2. Secondary Outcome: Survival
Description: To evaluate the progression-free survival and event-free survival in patients who receive therapy with fludarabine, Velcade, and rituximab.
Time Frame: 6 months
Population: Data for this secondary objective was not collected or analyzed due to the termination of the study.
Arm/Group | Fludarabine, Velcade and Rituximab
Number analyzed (Participants) | 0

3. Secondary Outcome: Toxicity
Description: To evaluate the toxicity profile of this regimen. Adverse event counts by grade are presented.
Time Frame: 6 months
Measure: Number; unit: number of adverse events
Arm/Group | Fludarabine, Velcade and Rituximab
Number analyzed (Participants) | 4
number of adverse events
  Total Adverse Events | 122
  Grade 1 Adverse Events | 77
  Grade 2 Adverse Events | 35
  Grade 3 Adverse Events | 9
  Grade 4 Adverse Events | 1
  Grade 5 Adverse Events | 0

4. Secondary Outcome: Biologic Interaction
Description: To explore the biologic interaction between fludarabine and Velcade and determine if Velcade can potentiate the DNA-damaging effect of fludarabine.
Time Frame: 6 months
Population: Data for this secondary objective was not collected or analyzed due to the termination of the study.
Arm/Group | Fludarabine, Velcade and Rituximab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Fludarabine, Velcade and Rituximab
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fludarabine, Velcade and Rituximab (N=4)
BLOOD/BONE MARROW - OTHER (SPECIFY, __) (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fludarabine, Velcade and Rituximab (N=4)
ALLERGIC REACTION/HYPERSENSITIVITY (INCLUDING DRUG FEVER) (Immune system disorders) | 1 (1)
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 1 (1)
ANOREXIA (Gastrointestinal disorders) | 1 (2)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 1 (1)
ATAXIA (INCOORDINATION) (Nervous system disorders) | 1 (1)
BRUISING (IN ABSENCE OF GRADE 3 OR 4 THROMBOCYTOPENIA) (Skin and subcutaneous tissue disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 3 (12)
CONSTITUTIONAL SYMPTOMS (General disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CREATININE (Investigations) | 1 (3)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 3 (6)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 4 (14)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 1 (1)
GASTRITIS (INCLUDING BILE REFLUX GASTRITIS) (Gastrointestinal disorders) | 1 (1)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 2 (3)
HEMOGLOBIN (Blood and lymphatic system disorders) | 3 (6)
HICCOUGHS (HICCUPS, SINGULTUS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HYPERTENSION (Cardiac disorders) | 1 (1)
INFECTION - OTHER (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / UPPER AERODIGESTIVE NOS (Infections and infestations) | 1 (1)
LEUKOCYTES (TOTAL WBC) (Blood and lymphatic system disorders) | 1 (1)
LEUKOENCEPHALOPATHY (RADIOGRAPHIC FINDINGS) (Nervous system disorders) | 1 (1)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 (7)
MAGNESIUM, SERUM-HIGH (HYPERMAGNESEMIA) (Investigations) | 1 (2)
MOOD ALTERATION / AGITATION (Psychiatric disorders) | 1 (1)
MOOD ALTERATION / ANXIETY (Psychiatric disorders) | 2 (2)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) / ORAL CAVITY (Surgical and medical procedures) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 2 (8)
NEUROPATHY: MOTOR (Nervous system disorders) | 1 (1)
NEUROPATHY: SENSORY (Nervous system disorders) | 2 (10)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Blood and lymphatic system disorders) | 1 (4)
NYSTAGMUS (Eye disorders) | 1 (1)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 1 (1)
PAIN / BACK (General disorders) | 1 (1)
PAIN / EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 1 (2)
PAIN / HEAD/HEADACHE (General disorders) | 1 (2)
PAIN / JOINT (Musculoskeletal and connective tissue disorders) | 1 (2)
PAIN / LYMPH NODE (Blood and lymphatic system disorders) | 1 (1)
PAIN - OTHER (General disorders) | 1 (1)
PLATELETS (Blood and lymphatic system disorders) | 3 (6)
RIGORS/CHILLS (General disorders) | 2 (4)
SEXUAL/REPRODUCTIVE FUNCTION - OTHER (Reproductive system and breast disorders) | 1 (1)
SWEATING (DIAPHORESIS) (General disorders) | 1 (1)
WATERY EYE (EPIPHORA, TEARING) (Eye disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This trial was terminated after accruing four subjects to do slow accrual. Sufficient data was not collected to complete the primary objective.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No